CLINICAL TRIAL: NCT03250715
Title: Effects of Low Level Laser Therapy on Functional Capacity and DNA Damage of Patients With Chronic Kidney Failure on Hemodialysis: Randomized Clinical Trial
Brief Title: Effects of Low Level Laser Therapy on Functional Capacity and DNA Damage of Patients With Chronic Kidney Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LLLT_CKF_HD
Record Dates: First submitted 2017-08-07; First posted 2017-08-16 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Low-Level Light Therapy; Renal Insufficiency, Chronic; Renal Dialysis; Clinical Trial
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Level Laser Therapy group (Experimental): Six points of application will be defined in the quadriceps and two points of application in the gastrocnemius. The parameters adopted for the irradiation will be: 30 Joules per application point, wavelength of 660 and 850 nm and output power of 200 mW. Each point will be radiated for 30 seconds.
  Interventions: Other: Low Level Laser Therapy
- Control group (No Intervention): This group will receive no intervention. This group will be evaluated before the intervention, after four and eight weeks of follow up.

INTERVENTIONS:
Other: Low Level Laser Therapy — For application of the LLLT in the quadriceps muscle the patient will be in dorsal decubitus, with the legs extended and will be defined by the palpation of the muscle belts six points of application: two points in the distal region of the vastus medialis muscle, two points of the distal region of the vastus lateral muscle and two points of the central region of the rectus femoris muscle. For the application of LLLT in the gastrocnemius muscle the patient will remain in the supine position, but will be oriented to keep the hips and knees flexed at 90º and 45º respectively. Two application points will be defined, one in the lateral ventricle and the other in the medial ventricle, but both in the distal region of the muscle.
  Other Names: Low-Level Light Therapy
  Arms: Low Level Laser Therapy group

SUMMARY:
This study aims to verify the effects of low level laser therapy (LLLT) on functional capacity, DNA damage, lower limbs muscle strength, quadriceps muscle architecture, muscle pain and perception of lower limb fatigue, inflammatory profile, oxidative stress and quality of life of patients with chronic kidney failure on hemodialysis. Patients will be randomized into two groups: the control group and the LLLT group. The control group will only be evaluated and reassessed. The LLLT group in addition to the evaluations will receive LLLT three times a week for eight weeks during HD. The evaluations will be performed pre-intervention, after 4 and 8 weeks of therapy. However, the muscle architecture evaluation will be performed only at pre intervention and after 8 weeks.

The evaluations carried out are: six-minute walk test for functional capacity; alkaline comet assay for DNA damage; sit-and-lift test, and load cell dynamometry for evaluation of lower limbs muscle strength; quadriceps ultrasonography for muscle architecture and echogenicity; visual analogue scale for pain; subjective perception of effort by Borg scale for fatigue; measurement of interleukins 6 and 10, tumor necrosis factor, reative C protein and muscle damage markers (lactate, creatine kinase) for the inflammatory profile; protein carbonylation, superoxide dismutase, catalase, total sulfuric acid and dichlorofluorescein diacetate for oxidative stress and application of the Kidney Disease and Quality-of-Life-Short-Form and EQ-5D questionnaires for quality of life.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) consists of kidney damage and progressive and irreversible loss of kidney function and in its later stage (terminal phase) is called chronic kidney failure (CKF). Although hemodialysis (HD) substitutes some of the lost renal functions, patients suffer from some changes that characterize uremic syndrome, such as peripheral motor neuropathy, osteomalacia, cardiac and musculoskeletal myopathies, anemia, among other alterations.

This study aims to verify the effects of low level laser therapy (LLLT) on functional capacity, DNA damage, lower limbs muscle strength, quadriceps muscle architecture, muscle pain and perception of lower limb fatigue, inflammatory profile, oxidative stress and quality of life of patients with chronic kidney failure on hemodialysis. Patients will be randomized into two groups: the control group and the LLLT group. The control group will only be evaluated and reassessed. The LLLT group in addition to the evaluations will receive LLLT three times a week for eight weeks during HD. The evaluations will be performed pre-intervention, after 4 and 8 weeks of therapy. However, the muscle architecture evaluation will be performed only at pre intervention and after 8 weeks.

The evaluations carried out are: a six-minute walk test for functional capacity; alkaline comet assay for DNA damage; sit-and-lift test, and load cell dynamometry for evaluation of lower limbs muscle strength; quadriceps ultrasonography for muscle architecture and echogenicity; visual analogue scale for pain; subjective perception of effort by Borg scale for fatigue; measurement of interleukins 6 and 10, tumor necrosis factor, reative C protein and muscle damage markers (lactate, creatine kinase) for the inflammatory profile; protein carbonylation, superoxide dismutase, catalase, total sulfuric acid and dichlorofluorescein diacetate for oxidative stress and application of the Kidney Disease and Quality-of-Life-Short-Form and EQ-5D questionnaires for quality of life.

The expected results at the end of the protocol are: greater distance covered in the walking test; reduction of DNA damage, increase in lower limbs strength; maintenance of muscle mass; reduction of pain and fatigue levels as well as the inflammatory profile and levels of oxidative stress, as well as improvement in the quality of life for the group LLLT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney failure on hemodialysis for more than 3 months;
* Dialysis with weekly frequency of 3 times/week;
* Adequate urea clearance rate during hemodialysis (Kt/V ≥ 1.2 or URR ≥65%).

Exclusion Criteria:

* Cognitive dysfunction
* Epidermal lesions at the site of laser application
* Patients with active carcinoma
* Patients with recent sequel of stroke (three months)
* Recent myocardium acute infarction (two months)
* Uncontrolled hypertension (SBP> 230 mmHg and DBP> 120 mmHg)
* Grade IV heart failure according to the New York Heart Association or decompensated
* Unstable angina
* Peripheral vascular changes in lower limbs such as deep venous thrombosis
* Disabling osteoarticular or musculoskeletal disease
* Uncontrolled diabetes (glycemia> 300mg/dL)
* Febrile condition and/or infectious disease
* Active smoking.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Functional Capacity | Before intervention, after 4 and 8 weeks
  Functional capacity will be assessed by the Six-Minute Walk Test
Change in DNA Damage | Before intervention, after 4 and 8 weeks
  DNA damage will be assessed by the alkaline comet assay

SECONDARY OUTCOMES:
Change in Muscle Strength of Lower Limbs | Before intervention, after 4 and 8 weeks
  Muscle strength of lower limbs will be assessed by dynamometry
Change in Muscle Architecture | Before intervention and after 8 weeks
  Muscle architecture of quadriceps will be assessed by ultrasonography
Change in Muscle Pain | Before intervention, after 4 and 8 weeks
  Muscle pain will be assessed by analogic visual scale
Change in Fatigue of Lower Limbs Fatigue of lower limbs | Before intervention, after 4 and 8 weeks
  Fatigue of lower limbs will be assessed by Borg's subjective effort perception scale Fatigue of lower limbs will be assessed by Borg's effort perception scale
Change in Oxidative Stress | Before intervention, after 4 and 8 weeks
  Oxidative stress will be assessed by measurement of oxidative and antioxidant markers
Change in Inflammatory Profile | Before intervention, after 4 and 8 weeks
  Inflammatory profile will be assessed by measurement of interleukins and markers of muscle damage
Change in Quality of Life | Before intervention and after 8 weeks
  Quality of life will be assessed by Kidney Disease and Quality-of-Life Short-Form questionnaire
Change in Quality of Life | Before intervention, after 4 and after 8 weeks
  Quality of life will be assessed by EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided